CLINICAL TRIAL: NCT03115489
Title: Efficacy of Ketamine Infusion Compared With Traditional Anti-epileptic Agents in Refractory Status Epilepticus- a Pilot Study
Brief Title: Efficacy of Ketamine Infusion Compared With Traditional Anti-epileptic Agents in Refractory Status Epilepticus
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low eligibility of patients, no successful recruitment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Vinodkumar Singh, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F151214004
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Refractory Epilepsy
Keywords: seizure; glutamate activation; N-Methyl D-Aspartate; gamma-aminobutyric acid receptor; Ketamine
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures | interventions — Sensitivity Training Groups; Benzodiazepines; Barbiturates; Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Traditional Treatment (Group T) (Placebo Comparator): Group T patients will be placed into burst suppression with the traditional drug infusions which include any single or combination of drugs; usually benzodiazepines, barbiturates and or propofol.
  Interventions: Drug: Traditional Treatment (Group T)
- Ketamine Infusion (Group K) (Active Comparator): Patients in the group K arm will receive a loading dose of 2.5 mg/kg of ketamine followed by a continuous infusion with a starting dose of 3mg/kg/hr with titration in 1mg/kg/hr increments until burst suppression is achieved or a maximum dose of 10mg/kg/hr is reached. After 48 hours of burst suppression the ketamine dosage will be reduced by 2mg/kg/hr in a stepwise fashion to evaluated for EEG or clinical evidence of seizure recurrence.
  Interventions: Drug: Ketamine Infusion (Group K)

INTERVENTIONS:
Drug: Traditional Treatment (Group T) — Patients will receive traditional drug infusions
  Other Names: benzodiazepines, barbiturates, propofol
  Arms: Traditional Treatment (Group T)
Drug: Ketamine Infusion (Group K) — Patients will receive loading dose of 2.5 mg/kg of ketamine followed by a continuous infusion with a starting dose of 3mg/kg/hr with titration in 1mg/kg/hr increments until burst suppression is achieved or a maximum dose of 10mg/kg/hr is reached
  Other Names: Ketalar
  Arms: Ketamine Infusion (Group K)

SUMMARY:
The study will investigate the efficacy of the N-methyl-D-aspartate receptor antagonist ketamine as a first line agent in refractory status epilepticus versus traditional general anesthetic agents used for burst suppression that target the gamma-aminobutyric acid adrenergic receptors.

DETAILED DESCRIPTION:
The traditional treatment for refractory status epilepticus includes diazepam, midazolam, valproic acid, thiopental and propofol. These medications fail to control seizure activity in 20-40% of patients. This is attributed to decrease in activity of gamma-aminobutyric acid receptors along with reciprocal up regulation of N-Methyl-D-aspartate receptors. Glutamate activation of N-methyl-D-aspartate receptors promotes calcium influx and excitotoxicity. Ketamine, an intravenous anesthetic agent which is a non-competitive antagonist of N-methyl-D-aspartate receptors can block the flow of Ca and Na and by combining with phencyclidine binding sites inside the ion channel of N-methyl-D-aspartate receptors, reduce the epileptiform burst discharges and after potential. Therefore, targeting the N-methyl-D-aspartate receptors with ketamine may provide a novel approach to control refractory seizures. Moreover, by blocking glutamate mediated N-methyl-D-aspartate receptor induced neurotoxicity, ketamine may render neuroprotection. Ketamine also provides additional advantage of hemodynamic stability. Currently, ketamine is used as a last resort drug in the treatment of refractory status epilepticus.

The specific aim is to determine whether continuous infusion of ketamine as a first line agent for refractory status epilepticus is effective in controlling seizures.

The central hypothesis of our proposal is that early treatment with ketamine will be much more efficacious in controlling refractory status compared to the traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years of age with a diagnosis of status epilepticus
* Considered for burst suppression therapy after failing 2 or 3 anti-epileptic medications

Exclusion Criteria:

* Post anoxic status epilepticus
* Pregnant women, as confirmed by urine, or blood human chorionic gonadotropin, ultrasound or physical exam
* Prisoners
* Age less than 18 years
* Allergy or sensitivity to the drug in question

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Time taken for burst suppression | Baseline to 1 hr
  Average time for burst suppression
Time taken for termination of seizures | Baseline to 24 hrs
  Average time for seizures to terminate

SECONDARY OUTCOMES:
Use of vasopressors | baseline to 72 hrs
  The need of vasopressors
Number of days on ventilator | Baseline to 72 hrs
  Total number of days patient is on the ventilator
Length of stay in ICU | Baseline to 72 hrs postoperatively
  Total number of days in the ICU
Use of parenteral or enteral nutrition | Baseline to 72 hrs postoperatively
  Nutrition provided through a feeding tube or catheter
Medical imaging results | Post-op Day 2 to Post-op day 10
  MRI scans 7 to 10 days after burst suppression
Mortality | baseline to post-op day 10
  death

CONTACTS AND LOCATIONS:
Overall Officials: Vinodkumar Singh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosati A, De Masi S, Guerrini R. Ketamine for Refractory Status Epilepticus: A Systematic Review. CNS Drugs. 2018 Nov;32(11):997-1009. doi: 10.1007/s40263-018-0569-6. PMID 30232735